CLINICAL TRIAL: NCT00535678
Title: A Multicenter Study to Test Digital Breast Tomosynthesis (DBT) Compared to Full-Field Digital Mammography (FFDM) in Detecting Breast Cancer. Part 1. Women Undergoing Screening Mammography
Brief Title: Testing Digital Breast Tomosynthesis vs. Regular Mammogram in Detecting Breast Cancer in Women Having Screening Mammogram
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: GE Healthcare - Kevin Horgan, GE Healthcare
Other Study IDs: GE 190-001
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-04

CONDITIONS: Breast Cancer
Keywords: Mammography; mammogram; breast; Abnormal and normal breast tissue
MeSH Terms: conditions — Breast Neoplasms; Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To compare DBT and FFDM for screening effectiveness in women who present for screening mammography with respect to screening recall rate.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years or older for screening mammography
* Able and willing to comply with study procedures, and have signed and dated the informed consent form
* The subject is surgically sterile or postmenopausal

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Has signs or symptoms of breast cancer
* Has been previously included in this study
* Has breast implants
* Has a history of breast cancer and is in active treatment
* Has breasts too large to be adequately positioned for the DBT examination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women referred for normal screening mammogram
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Compare the diagnostic performance of FFDM and DBT in detecting and excluding breast cancer in asymptomatic women.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Longcore, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States